CLINICAL TRIAL: NCT03219905
Title: Does "Kinesio-taping" Affect Standing Balance in Healthy Individuals? A Randomized Controlled Pilot Trial
Brief Title: Does "Kinesio-taping" Affect Balance in Healthy Individuals?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Haydar Gok, Professor of Physical Medicine and Rehabilitation, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-213-14
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Balance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio-taping Group (Experimental): Therapeutic Kinesio-taping
  Interventions: Device: Therapeutic Kinesio-taping
- Control Group (Sham Comparator): Sham Kinesio-taping
  Interventions: Device: Sham Kinesio-taping

INTERVENTIONS:
Device: Therapeutic Kinesio-taping — The experimental group received a therapeutic Kinesio Tape application. Three "I" strips were applied to the both ankle joints for joint stability with subject's ankle at 90 degrees.
  Arms: Kinesio-taping Group
Device: Sham Kinesio-taping — The control group received a sham Kinesio Tape application. Ankle position was hold at minimally plantar flexion during taping. A"I" strip was placed from the anterior midfoot, not stretched and attached to the midline of anterior leg.
  Arms: Control Group

SUMMARY:
Kinesio-taping (KT) has recently gained so much popularity and a growing number of physicians started using it to alleviate musculoskeletal symptoms. It was originally developed by Kenzo Kase in 1976. The effects of KT on ankle proprioception and stability have been investigated in previous studies. However, these studies are limited and the current data is conflicting. Repeated application of KT in a patient with chronic ankle instability has been shown to be effective in improving balance. In basketball players with chronic ankle sprain, KT did not improve or inhibit balance. Application of KT did not cause a significant change in balance of healthy subjects. The aim of this study was to evaluate the immediate and short-term effects of KT on balance of healthy subjects.

DETAILED DESCRIPTION:
Thirty male healthy volunteers (between 18-40 ages) were screened for eligibility by physical examination and history. Informed written consent was obtained from all participants before enrollment. The research proposal was reviewed and approved by the Faculty Ethics Committee(No: 05-213-14).

This is a randomized sham controlled, double-blind pilot clinical trial. The block randomization method with a block size of 4 was used in order to allocate the subjects equally into two groups; Kinesiotaping (KT) and sham (control).To conceal the randomization sequence an independent researcher (HG) who is unaware of the baseline data carried out the procedure using a computer software. The researcher (MO) who was blinded to the allocationprocedure did the balance testing of all subjects, before (t0), immediately after (t1) and 24 hours after the application of KT (T2). The subjects were also blinded to the type of intervention.

Standard 2-inch (5-cm) Kinesio® Tex (Kinesio Holding Corporation, Albuquerque, NM) Tape was used for all applications in both groups. A certified KT practitioner (BST) did the all taping procedures. KT was applied bilaterally to the ankle joints. To ensure blinding of the assessor (MÖ), taping procedure was done in a separate room and subjects wore their socks after the application. The tape remained in place for 24 hours duration and subjects were instructed to participate in their normal daily activities, except shower.

The experimental group received a standardized therapeutic Kinesio Tape application. Three "I" strips were applied to the both ankle joints for joint stability with subject's ankle at 90 degrees. KT was applied according to the procedures recommended by the website of http://www.kttapeeurope.com/How-to-tape-Ankle-Stability (last accessed on July 7th, 2017). First strip was anchored 5 cm above the ankle. Then tape was applied down the outer ankle, across the bottom of the heel, and up the inner side of the ankle. The last 5cm of tape was laid without stretch. Second strip was anchored along the instep of the foot. Then tape was laid around the back of the heel and across the arch with 50% stretch. The last part of tape was laid down without stretch on inside of foot. Third strip was anchored same style along the outside of the foot. The tape was laid the around the back of the heel and across the arch with 50% stretch. The last 5 cm of the tape was laid down without stretch on insideof foot. The control group received a sham Kinesio Tape application. Ankle position was hold at minimally plantar flexion during taping. A"I" strip was placed from the anterior midfoot, not stretched and attached to the midline of anterior leg.

Each participant's height and weight were recorded and body mass index (BMI) was calculated. Balance measurements were made with a stabilometer, BiodexTM Balance System. A dynamic postural stability test was performed in a double-leg standing position with eyes open. Each test included three trials that lasted 20 seconds with a 10-second rest period between them. A mean score was calculated from three trials. Subjects were given a practice trial lasting 20 sec. to familiarize with the test. During the dynamic postural stability test three indices were calculated; (1) anteroposterior stability index (APSI), (2) mediolateral stability index (MLSI), (3) overall stability index (OSI). The OSI indicates the total variation in plate deviation (sway) from the horizontal plane. The APSI and MLSI indicate the deviation of the plate (sway) from the horizontal position in the sagittal and frontal planes, respectively. Since the values obtained during measurements indicate the amount of sway from the horizontal position, lower scores show better balance.

Non-parametric tests have been used due to the small sample size and skewed data distribution. The baseline demographic characteristics of the patients in each group were compared by Mann Whitney U test. The two-way mixed ANOVA was used to compare the mean differences between independent groups over time and to understand if there is an interaction between time and group factors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Age between 18-40 years
* polyneuropathy or neurological deficits

Exclusion Criteria:

Individuals with;

* lower extremity fractures
* knee or ankle ligamentous injury
* conditions affecting balance, knee, hip or spinal osteoarthritis
* lower extremity or back surgery
* polyneuropathy or neurological deficits

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mediolateral stability index (MLSI) | Change from Baseline in MLSI immediately after KT application
  A dynamic postural stability test which is performed in a double-leg standing position with eyes open.
Mediolateral stability index (MLSI) | Change from Baseline in MLSI 24 hours after KT application
  A dynamic postural stability test which is performed in a double-leg standing position with eyes open.

SECONDARY OUTCOMES:
Anteroposterior stability index (APSI) | Change from Baseline in APSI immediately after KT application
  A dynamic postural stability test which is performed in a double-leg standing position with eyes open.
Anteroposterior stability index (APSI) | Change from Baseline in APSI 24 hours after KT application
  A dynamic postural stability test which is performed in a double-leg standing position with eyes open.
Overall stability index (OSI) | Change from Baseline in OSI immediately after KT application
  A dynamic postural stability test which is performed in a double-leg standing position with eyes open.
Overall stability index (OSI) | Change from Baseline in OSI 24 hours after KT application
  A dynamic postural stability test which is performed in a double-leg standing position with eyes open.

CONTACTS AND LOCATIONS:
Overall Officials: Haydar Gok, Professor, Principal Investigator — Ankara University

REFERENCES:
- [Background] Wikstrom EA, Tillman MD, Kline KJ, Borsa PA. Gender and limb differences in dynamic postural stability during landing. Clin J Sport Med. 2006 Jul;16(4):311-5. doi: 10.1097/00042752-200607000-00005. PMID 16858214
- [Background] Gabriel RC, Abrantes J, Granata K, Bulas-Cruz J, Melo-Pinto P, Filipe V. Dynamic joint stiffness of the ankle during walking: gender-related differences. Phys Ther Sport. 2008 Feb;9(1):16-24. doi: 10.1016/j.ptsp.2007.08.002. Epub 2007 Sep 29. PMID 19083700
- [Background] Akbari A, Sarmadi A, Zafardanesh P. The effect of ankle taping and balance exercises on postural stability indices in healthy women. J Phys Ther Sci. 2014 May;26(5):763-9. doi: 10.1589/jpts.26.763. Epub 2014 May 29. PMID 24926148
- [Background] Tamburella F, Scivoletto G, Molinari M. Somatosensory inputs by application of KinesioTaping: effects on spasticity, balance, and gait in chronic spinal cord injury. Front Hum Neurosci. 2014 May 30;8:367. doi: 10.3389/fnhum.2014.00367. eCollection 2014. PMID 24910607
- [Background] Cortesi M, Cattaneo D, Jonsdottir J. Effect of kinesio taping on standing balance in subjects with multiple sclerosis: A pilot study\m1. NeuroRehabilitation. 2011;28(4):365-72. doi: 10.3233/NRE-2011-0665. PMID 21725170
- [Background] Kinzey SJ, Ingersoll CD, Knight KL. The effects of selected ankle appliances on postural control. J Athl Train. 1997 Oct;32(4):300-3. PMID 16558462
- [Background] Nunes GS, de Noronha M, Cunha HS, Ruschel C, Borges NG Jr. Effect of kinesio taping on jumping and balance in athletes: a crossover randomized controlled trial. J Strength Cond Res. 2013 Nov;27(11):3183-9. doi: 10.1519/JSC.0b013e31828a2c17. PMID 23439339
- [Background] Shields CA, Needle AR, Rose WC, Swanik CB, Kaminski TW. Effect of elastic taping on postural control deficits in subjects with healthy ankles, copers, and individuals with functional ankle instability. Foot Ankle Int. 2013 Oct;34(10):1427-35. doi: 10.1177/1071100713491076. Epub 2013 May 29. PMID 23720530
- [Background] Nakajima MA, Baldridge C. The effect of kinesio(R) tape on vertical jump and dynamic postural control. Int J Sports Phys Ther. 2013 Aug;8(4):393-406. PMID 24175126
- [Background] You SH, Granata KP, Bunker LK. Effects of circumferential ankle pressure on ankle proprioception, stiffness, and postural stability: a preliminary investigation. J Orthop Sports Phys Ther. 2004 Aug;34(8):449-60. doi: 10.2519/jospt.2004.34.8.449. PMID 15373008